CLINICAL TRIAL: NCT06676722
Title: A Prospective, Single-Arm, Exploratory Study of SBRT Combined With Nimotuzumab and Sequential Tislelizumab for Oligoprogressive Distant Recurrent/Metastatic Nasopharyngeal Carcinoma After Failure of First-Line Immunotherapy
Brief Title: SBRT Combined With Nimotuzumab and Tislelizumab for Oligoprogressive Recurrent/Metastatic Nasopharyngeal Carcinoma After Failure of Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, San-Gang Wu, Dr., The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023152
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Nasopharyngeal Cancinoma (NPC); SBRT; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): SBRT combined with Nimotuzumab followed by Tislelizumab
  Interventions: Drug: SBRT combined with Nimotuzumab followed by Tislelizumab

INTERVENTIONS:
Drug: SBRT combined with Nimotuzumab followed by Tislelizumab — BRT combined with 3 cycles of Nimotuzumab 400mg qw followed by maintain Tislelizumab for 2 years or until disease progression

SUMMARY:
This study is a single-arm, open-label, prospective, and exploratory investigation aimed at examining the short-term efficacy, specifically the objective response rate (ORR), of SBRT combined with Nimotuzumab followed by Tislelizumab in patients with recurrent/metastatic nasopharyngeal carcinoma who have experienced oligoprogression (1-5 metastatic lesions) after immunotherapy.

ELIGIBILITY:
1. Inclusion Criteria:

   1.1. Pathologically confirmed non-keratinizing nasopharyngeal carcinoma; 1.2. Patients with recurrent/metastatic nasopharyngeal carcinoma who have previously received first-line treatment including anti-PD-1 immune checkpoint inhibitor therapy and failed, presenting with oligoprogression (1-5 metastatic lesions); 1.3. Eligible to receive SBRT, Tislelizumab, and Nimotuzumab; 1.4. No history of other malignant tumors; 1.5. Male or female, aged 18-75 years; 1.6. Liver function: Total bilirubin ≤ Upper Limit of Normal (ULN); AST and ALT ≤ 2.5 × ULN; Alkaline phosphatase ≤ 5 × ULN; 1.7. Renal function: Creatinine clearance ≥ 80 mL/min; 1.8. Hematological tests: Absolute neutrophil count (ANC) ≥ 2 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL; 1.9. No severe dysfunction of heart, lung, and other vital organs; 1.10. Performance Status (PS) score ≤ 2.
2. Exclusion Criteria:

2.1. Disagree to sign the informed consent form; 2.2. Patients who cannot comply with regular follow-ups due to psychological, social, family, or geographical reasons; 2.3. Receiving other experimental treatments as part of a clinical study (during the treatment period of the clinical study); 2.4. Severe, uncontrolled infections or medical conditions; 2.5. Major organ dysfunction, decompensated heart, lung, kidney, or liver failure, unable to tolerate radiotherapy or immunotherapy; 2.6. Factors affecting drug administration, distribution, metabolism, or excretion, such as mental abnormalities, central nervous system abnormalities, chronic diarrhea, ascites, pleural effusion, etc.; 2.7. Overexposure to glucocorticoids within 2 weeks before immunotherapy; 2.8. Long-term use of immunosuppressive agents after organ transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR） | 6 months
  To investigate the short-term efficacy, specifically the objective response rate (ORR), of SBRT combined with Nimotuzumab followed by Tislelizumab in patients with recurrent/metastatic nasopharyngeal carcinoma who have experienced oligoprogression (1-5 metastatic lesions) after immunotherapy.

SECONDARY OUTCOMES:
Progression-free survival rate | 6 months
  The proportion of patients who are alive and free of disease relapse at 6 months after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No